CLINICAL TRIAL: NCT01413555
Title: Multicenter Implementation of a Quality Improvement Program to Reduce Blood Culture Contamination in the Emergency Department
Brief Title: Multicenter Blood Culture Quality Improvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Community Health Network (Other); C. R. Bard (Industry)
Responsible Party: Principal Investigator, Wesley Self, Asst Professor, Department of Emergency Medicine, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VHRPP - 101722
Record Dates: First submitted 2011-08-08; First posted 2011-08-10 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Bacteremia
Keywords: blood culture; emergency department; quality improvement
MeSH Terms: conditions — Bacteremia; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood Culture QI Program (Experimental)
  Interventions: Other: Blood Culture QI Program

INTERVENTIONS:
Other: Blood Culture QI Program — The Blood Culture QI Program contains four components:(1) education: content knowledge and standardized experiential training on sterile technique designed for ED nurses; (2) process redesign: conversion of blood culture collection from a clean to a sterile technique using the Blood Culture Sterile Kit; (3) a checklist outlining optimal use of the Kit; (4) feedback of blood culture contamination rates to ED nurses who collect them.
  Other Names: ChloraPrep

SUMMARY:
False positive blood culture results due to specimen contamination with bacteria inhabiting patients' skin is a common problem in emergency departments (EDs) in the United States. Contaminated blood cultures lead to patient harm through unnecessary hospitalizations and ED visits, delays in surgery, unneeded antibiotics, and unnecessary procedures. The investigators have developed a multifaceted quality improvement improvement bundle (The Blood Culture QI Program) designed to minimize blood culture contamination in the ED. In this study, the investigators will implement the quality improvement bundle in six community hospital EDs and evaluate its effectiveness at reducing contamination.

DETAILED DESCRIPTION:
The Blood Culture QI Program has four components: (1) education: content knowledge and standardized experiential training on sterile technique designed for ED nurses; (2) process redesign: change in patient safety attitude and conversion of blood culture collection from a clean to a sterile technique; (3) checklist use: reinforcement of optimal blood culture collection technique at the point of care; (4) feedback: systematic charting and reporting of contamination rates to the ED nurses who collect cultures. In order to convert blood culture collection into a fully sterile procedure, the investigators developed the Sterile Blood Culture Collection Kit, a novel materials kit that contains the equipment needed to collect a culture using sterile technique, including: (1) a 3ml solution of 2% chlorhexidine gluconate - 70% isopropyl alcohol (Chloraprep, CareFusion) skin prep device; (2) a sterile drape; (3) a sterile needle; and (4) gauze.

The investigators will evaluate the effectiveness of the Blood Culture QI Program after implementing it in six community hospital EDs. Our study will compromise six replications of an interrupted time series study wherein each replication will be powered for internal validity to test the hypothesis of decreasing the contamination rate by 50% at each site. A stepped wedge (also called multiple baseline) design will be used to implement the program across hospitals to evaluate the generalizability (external validity) of program effectiveness. The primary analysis will be an interrupted time series analysis at each site comparing the proportion of ED blood cultures contaminated during a post-implementation intervention period with a pre-intervention baseline period.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a blood culture ordered for clinical purposes in one of the participating centers during the study period.

Exclusion Criteria:

* Age < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14889 (Actual)
Dates: Start 2011-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Biweekly proportion of ED blood cultures contaminated | 1 year
  In an interrupted time series design, we will compare the proportion of blood cultures contaminated during an intervention period after the implementation of the Blood Culture QI Program to a baseline period before implementation. We will complete six separate interrupted time series analyses with one at each of six hospitals. The intervention and baseline period duration will be approximately one year at each hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Wesley H. Self, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (2):
- United States (2):
  - Vanderbilt Emergency Medicine, Nashville, Tennessee
  - Vanderbilt University Medical Center Emergency Medicine, Nashville, Tennessee

REFERENCES:
- [Background] Archibald LK, Pallangyo K, Kazembe P, Reller LB. Blood culture contamination in Tanzania, Malawi, and the United States: a microbiological tale of three cities. J Clin Microbiol. 2006 Dec;44(12):4425-9. doi: 10.1128/JCM.01215-06. Epub 2006 Oct 4. PMID 17021063
- [Background] Norberg A, Christopher NC, Ramundo ML, Bower JR, Berman SA. Contamination rates of blood cultures obtained by dedicated phlebotomy vs intravenous catheter. JAMA. 2003 Feb 12;289(6):726-9. doi: 10.1001/jama.289.6.726. PMID 12585951
- [Background] Qamruddin A, Khanna N, Orr D. Peripheral blood culture contamination in adults and venepuncture technique: prospective cohort study. J Clin Pathol. 2008 Apr;61(4):509-13. doi: 10.1136/jcp.2007.047647. Epub 2007 Aug 30. PMID 17761739
- [Background] Bates DW, Goldman L, Lee TH. Contaminant blood cultures and resource utilization. The true consequences of false-positive results. JAMA. 1991 Jan 16;265(3):365-9. PMID 1984535
- [Background] Little JR, Murray PR, Traynor PS, Spitznagel E. A randomized trial of povidone-iodine compared with iodine tincture for venipuncture site disinfection: effects on rates of blood culture contamination. Am J Med. 1999 Aug;107(2):119-25. doi: 10.1016/s0002-9343(99)00197-7. PMID 10460041
- [Background] Gander RM, Byrd L, DeCrescenzo M, Hirany S, Bowen M, Baughman J. Impact of blood cultures drawn by phlebotomy on contamination rates and health care costs in a hospital emergency department. J Clin Microbiol. 2009 Apr;47(4):1021-4. doi: 10.1128/JCM.02162-08. Epub 2009 Jan 26. PMID 19171686
- [Background] Souvenir D, Anderson DE Jr, Palpant S, Mroch H, Askin S, Anderson J, Claridge J, Eiland J, Malone C, Garrison MW, Watson P, Campbell DM. Blood cultures positive for coagulase-negative staphylococci: antisepsis, pseudobacteremia, and therapy of patients. J Clin Microbiol. 1998 Jul;36(7):1923-6. doi: 10.1128/JCM.36.7.1923-1926.1998. PMID 9650937
- [Background] Zwang O, Albert RK. Analysis of strategies to improve cost effectiveness of blood cultures. J Hosp Med. 2006 Sep;1(5):272-6. doi: 10.1002/jhm.115. PMID 17219512